CLINICAL TRIAL: NCT01523678
Title: Phase II Study of Weekly Paclitaxel/Carboplatin in Combination With Prophylactic G-CSF in the Treatment of Gynaecological Cancers
Brief Title: Weekly Paclitaxel/Carboplatin With Neupogen in Gynaecological Cancers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Belgian Gynaecological Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BGOG-ov5; 2010-022482-95 (EudraCT Number)
Record Dates: First submitted 2012-01-24; First posted 2012-02-01 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Ovarian Cancer; Endometrial Cancer; Uterine Cervical Cancer
Keywords: Ovarian Cancer; Endometrial Cancer; Endometrial Carcinoma; Uterine Cervical Cancer; Paclitaxel; Carboplatin; Neupogen; Filgrastim; Ovarian Diseases; Peritoneal Diseases; Fallopian Tube Diseases; Endocrine System Diseases; Endometrial Diseases; Uterine Cervical Diseases; Neoplasms; Neoplasms, Glandular and Epithelial; Ovarian Neoplasms; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Neoplasms, Endometrial; Cervical Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Antineoplastic Agents, Phytogenic; Genital Diseases, Female
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms; Ovarian Diseases; Peritoneal Diseases; Fallopian Tube Diseases; Endocrine System Diseases; Uterine Diseases; Uterine Cervical Diseases; Neoplasms; Neoplasms, Glandular and Epithelial; Peritoneal Neoplasms; Fallopian Tube Neoplasms; Genital Neoplasms, Female; Urogenital Neoplasms; Genital Diseases, Female | interventions — Filgrastim; Paclitaxel; Carboplatin

ARMS (1):
- Filgrastim (Experimental)
  Interventions: Drug: Filgrastim; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Drug: Filgrastim — All subjects will receive standard treatment with paclitaxel followed by carboplatin intravenously during 18 weeks. Filgrastim (Neupogen) will be given prophylactically on day 5. An additional dose will be given on day 6 in case of severe neutropenia during the course of the trial.
Drug: Paclitaxel — All subjects will receive standard treatment with paclitaxel followed by carboplatin intravenously during 18 weeks. Filgrastim (Neupogen) will be given prophylactically on day 5. An additional dose will be given on day 6 in case of severe neutropenia during the course of the trial.
Drug: Carboplatin — All subjects will receive standard treatment with paclitaxel followed by carboplatin intravenously during 18 weeks. Filgrastim (Neupogen) will be given prophylactically on day 5. An additional dose will be given on day 6 in case of severe neutropenia during the course of the trial.

SUMMARY:
Rationale: The administration of prophylactic G-CSF may reduce the toxicity of a weekly paclitaxel/carboplatin regimen in gynaecological cancers.

Purpose: This multicenter phase II trial is studying the side effects of weekly paclitaxel/carboplatin when given with prophylactic G-SCF in patients with recurrent epithelial ovarian-, primary peritoneal or fallopian tube cancers, endometrial carcinoma or cervical carcinoma. Data obtained in this trial will be compared with historical data as published earlier.

The trial will include 3 cohorts of 36 patients:

* Subjects with ovarian, fallopian tube or peritoneal carcinoma
* Subjects with endometrial cancer
* Subjects with cervical carcinoma

Treatment:

Subjects will receive Paclitaxel 60 mg/m² followed by Carboplatin AUC 2.7 intravenously weekly during 18 weeks. Filgrastim (Neupogen) will be given to all patients on day 5 and possibly on day 6 of each course. Subjects will be evaluated by CT/MRI scan after 9 cycles of chemotherapy (week 10), after 18 cycles of chemotherapy, then every 6 months for the next 2 years and then if clinically indicated. Subjects who develop disease progression will discontinue therapy. Subjects who have no evidence of disease progression after completion of study therapy will be followed until disease progression, withdrawal of informed consent, or death.

DETAILED DESCRIPTION:
Primary objective:

- To evaluate the occurrence of grade 4 neutropenia during weekly paclitaxel/carboplatin with prophylactic G-CSF

Secondary objectives:

* To evaluate per cohort the occurrence of grade 4 neutropenia
* To evaluate other toxicities
* To evaluate the dose reductions or dose delays in the chemotherapy
* To determine the progression free survival according to RECIST v1.1
* To evaluate the response rate and overall survival

ELIGIBILITY:
Inclusion Criteria:

All cohorts:

* Female subjects more than 18 years of age
* Performance status must be ECOG 0-2.
* Adequate organ function
* Measurable disease by RECIST version 1.1 or CA125 progression according to the GCIG definition (Vergote et al).
* Written informed consent

Ovarian, fallopian tube or peritoneal carcinoma cohort:

* Histologically confirmed diagnosis of invasive epithelial ovarian,fallopian tube, or peritoneal carcinoma (serous, mucinous, endometrioid,clear cell, or carcinosarcomas are eligible).
* Patients should have received at least 1 earlier platin treatment but should be platin refractory (progression within 28 days after the last dose of platin) or platin resistant (progression within 6 months after last dose of platin therapy).
* Earlier weekly or dose-dense regimens with paclitaxel and carboplatin are not allowed. Consolidation after the last platin dose with non-platinum containing chemotherapy or molecular targeted drugs is allowed

Endometrial carcinoma cohort

* Histologically confirmed diagnosis of endometrial carcinoma (endometrioid,adenoacanthoma, adenosquamous, serous, clear cell carcinoma or carcinosarcomas are eligible).
* Recurrent or advanced endometrial carcinoma can be included.
* Earlier platin therapy is allowed. But earlier weekly or dose-dense regimens with paclitaxel and carboplatin are not allowed.

Cervical carcinoma cohort

* Histologically confirmed diagnosis of cervical carcinoma (adenocarcinoma or squamous carcinomas are eligible).
* Recurrent or advanced endometrial carcinoma can be included.
* Earlier platin (including concomitant with radiotherapy) therapy is allowed. But earlier weekly or dose-dense regimens with paclitaxel and carboplatin are not allowed.

Exclusion Criteria:

* Other histologies than those mentioned above such as non-epithelial ovarian carcinomas, neuro-endocrine tumors, sarcomas, metastases from other primary tumors, ...
* Earlier weekly or dose-dense paclitaxel and carboplatin regimen.
* Any unstable or serious condition e.g. uncontrolled infection requiring systemic therapy.
* Prior other malignancies treated primarily or for recurrence within 3 years prior to inclusion in this study, except for completely resected non- melanomatous skin carcinoma or successfully treated in situ carcinoma of the skin or cervix of the uterus.
* Any serious and/or unstable pre-existing medical, psychiatric, or other condition that could interfere with subject's safety, provision of informed consent, or compliance to study procedures
* Metastatic disease to the brain or leptomeninges.
* Treatment with any of the following anti-cancer therapies:
* radiation therapy, surgery or tumor embolization within 14 days prior to the first dose of study chemotherapy.
* chemotherapy, immunotherapy, biologic therapy, investigational therapy or hormonal therapy within 14 days or five half-lives of a drug (whichever is longer) prior to the first dose of study drug
* Known immediate or delayed hypersensitivity reaction or idiosyncrasy to drugs similar or related to Paclitaxel, Carboplatin or G-CSF.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2012-02; Primary Completion 2014-05 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Occurrence of grade 4 neutropenia | 2.5 years

SECONDARY OUTCOMES:
Occurence of other toxicities | 2.5 years
Occurence of dose reductions and dose delays | 2.5 years
Progression free survival | 3 years, 7 years
Overall survival | 3 years, 7 years

CONTACTS AND LOCATIONS:
Locations (17):
- Belgium (17):
  - Cliniques du Sud-Luxembourg, Arlon
  - Imeldaziekenhuis, Bonheiden
  - AZ Klina, Brasschaat
  - Grand Hôpital de Charleroi, Charleroi
  - St. Maarten Duffel, Duffel
  - UZ Antwerpen, Edegem
  - Jan Yperman Ziekenhuis, Ieper
  - AZ Groeninge, Kortrijk
  - CHU Tivoli, La Louvière
  - UZ Leuven, Leuven
  - Centre Hospitalier de l'Ardenne, Libramont
  - Centre Hospitalier Régional de la Citadelle, Liège
  - CHU Sart Tilman Liège, Liège
  - Cliniques et maternité St. Elizabeth, Namur
  - AZ Damiaan, Ostend
  - AZ Nikolaas, Sint-Niklaas
  - Cliniques universitaires UCL de Mont-Godinne, Yvoir

REFERENCES:
- See also: BGOG website — http://www.bgog.eu/